CLINICAL TRIAL: NCT02615951
Title: Characterization of B Regulatory (Breg) Cells in Healthy Subjects and in Rheumatoid Arthritis (RA)
Brief Title: Characterization of Breg Cells
Acronym: Breg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other); Institut de Génétique Moléculaire de Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9461
Record Dates: First submitted 2015-05-28; First posted 2015-11-26 (Estimated); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteers; Arthritis, Rheumatoid
Keywords: Regulatory B cells (Breg); Genes; Cell surface proteins; Nutrient transporters; Chemokine receptors
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Nutrient transporters study (Other): Blood sampling from 10 patients vith RA and 10 control patient for biological analysis and measure of nutrient transporters expression
  Interventions: Other: blood sampling
- Chemokine receptors study (Other): Blood sampling from 10 patients vith RA and 10 control patient for biological analysis and measure of chemokine receptors expression
  Interventions: Other: blood sampling
- Genes study (Other): Blood sampling from 10 patients vith RA and 10 control patient for biological analysis and measure of genes expression
  Interventions: Other: blood sampling
- Protein surface study (Other): Blood sampling from 10 patients vith RA and 10 control patient for biological analysis and measure of protein surface expression
  Interventions: Other: blood sampling
- Protein surface & genes data validation (Other): Blood sampling from 10 patients vith RA and 10 control patient for biological analysis and measure for validation of the data from "protein surface study" and "genes study" arms analysis.
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — Blood sample retrieval for biological and genetic analysis and comparison

SUMMARY:
Recently, it has been shown that B cells could also have regulatory functions through the secretion of interleukin 10 (IL-10). They are called the B regulatory cells (Breg). In the mouse model the most commonly used of rheumatoid arthritis, collagen-induced arthritis (CIA), the transfer Breg helps prevent the development of CIA and cure established arthritis. The investigators have recently shown that Breg were decreased in patients with RA compared to controls and that the rate of Breg was inversely correlated with disease activity and autoantibody. These results thus suggest that the lack of IL-10 secretion by B cells plays an important role in the pathophysiology of RA. Nevertheless, in humans, the Breg remain poorly understood. The main objective of this project is to better characterize the B capable of producing IL-10 both in subjects with RA and controls. Understanding which induces the secretion of IL-10 by B could allow to consider new therapeutic approaches in autoimmune diseases, including in RA.

The investigators therefore aim to identify nutrient transporters, chemokine receptors, genes and surface proteins differentially expressed between Breg and other B cells in patients with RA and in controls.

DETAILED DESCRIPTION:
Rational: Rheumatoid arthritis (RA), the most common inflammatory joint disease, is often associated with irreversible joint destruction and can involve the prognosis of patients. If treatments to stabilize the disease are now available, research continues to try to permanently cure the disease. It is well established that the B cells have a pathogenic role in RA. More recently, it has been shown that B cells could also have regulatory functions through the secretion of interleukin 10 (IL-10). They are called the B regulatory cells (Breg). In the mouse model the most commonly used of rheumatoid arthritis, collagen-induced arthritis (CIA), the transfer Breg helps prevent the development of CIA and cure established arthritis. The investigators have recently shown that Breg were decreased in patients with RA compared to controls and that the rate of Breg was inversely correlated with disease activity and autoantibody levels. These results thus suggest that the lack of IL-10 secretion by B cells plays an important role in the pathophysiology of RA. Nevertheless, in humans, the Breg remain poorly understood. The project's main objective is to better characterize the B capable of producing IL-10 both in subjects with RA and controls. Understanding which induces the secretion of IL-10 by B could allow to consider new therapeutic approaches in autoimmune diseases, including in RA.

Objectives:

Principal: To identify nutrient transporters and chemokine receptors differentially expressed between Breg and other B cells in patients with RA.

Secondary:

* To identify genes and surface proteins differentially expressed between Breg and other B Lymphocytes (BL) in patients with RA.
* To identify nutrient transporters, chemokine receptors, genes and surface proteins differentially expressed between Breg and other BL in healthy subjects.
* To compare the expression of nutrient transporters, chemokine receptors, genes and surface proteins between Breg Breg controls and subjects with RA.

Methods:

Design: Cross-sectional study involving bicentric rheumatology services in Montpellier and Nîmes to recruitment; our research team at the Translational IGMM Nîmes and immunology laboratory for biological analyzes.

Population:

* RA: patient meets the criteria ACR (American College of Rheumatology) -EULAR (European League Against Rheumatism) 2010, naïve and biotherapy with corticosteroids less than 10 mg / day, stable for at least a week.
* Controls: matched for age and sex to RA patients, with no systemic disease.

Endpoints

* Main: the average flow cytometry fluorescence intensity nutrient carriers and the percentage of BL expressing the different chemokine receptors
* Secondary: transcriptome analysis and proteomics surface with cytometric confirmation of protein expression of RNA and proteins identified.

Number of subjects: 50 controls and 50 RA patients (10 each for each of the 3 methods of comparison Breg / B IL10- and 10 each for each of the two stages of validation). Each patient will have a visit. The expected study duration is 2 years.

Statistical analysis: Comparing ratios B + IL-10 / IL-10-B between RA patients and controls by Student or Mann-Whitney tests.

Expected Results and Prospects: This project will allow us to better define and understand the Breg in patients with RA and in controls. If the investigators can find specific extracellular markers for Breg, this will simplify the further study of these cells. Understanding allowing BL becoming regulator and this explains the lack of IL-10 by the BL in RA could open new therapeutic perspectives.

ELIGIBILITY:
Inclusion Criteria:

* RA responding to ACR/EULAR 2010 criteria

Exclusion Criteria:

* steroid> 10 mg/d
* previous use of biological disease-modifying antirheumatic drug (DMARD)
* age<18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10-02 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Identification of nutrient transporters' and of chemokine receptors' differentially expressed between Breg and other B cells in patients with RA | after analysis of the blood sample from the subject selected for the primary outcome mesure. Estimated at half a year after subject recruitement started
  Comparison between Breg (B IL-10+) and IL-10 non secreting B lymphocytes (B IL-10 -) in RA patient of :
  * Medium fluorescence intensity of B lymphocytes for ASCT2, Glut1, PiT1, PiT2, RFT1&3
  * Percentage of B lymphocytes expressing chemokine receptors CCR4, CCR7, CCR9, CXCR3, CXCR4 and CXCR5

SECONDARY OUTCOMES:
Identification of genes and surface receptors expressed differentially between Breg and others B cells in patients with RA | Estimated at 6 month after end of subject recruitement
Identification of nutrient transporters and chemokine receptors expressed differentially between Breg and others B cells in control patients | Estimated at 6 month after end of subject recruitement
: Identification of genes and surface receptors expressed differentially between Breg and others B cells in control patients | Estimated at 6 month after end of subject recruitement
Comparison of nutrient transporters, chemokine receptors, gene and protein surface expression expressed between Breg in patients with RA and Breg in control patients | Estimated at 6 month after end of subject recruitement

CONTACTS AND LOCATIONS:
Overall Officials: Claire I Daien, MD PhD, Principal Investigator — Montpellier teaching hospital
Locations (1):
- Regional University Hospital, Montpellier, Hérault, France